CLINICAL TRIAL: NCT03792165
Title: Effects of Action Observation Therapy on Pain and Brain Hemodynamics in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Lecturer, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATADEK 2017/8
Record Dates: First submitted 2018-12-28; First posted 2019-01-03 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis; Action Observation Therapy; Functional Near Infared Spectroscopy; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation therapy and exercise (Experimental): Video of normal human movement and Strengthening and stretching exercises for hip and knee muscles
  Interventions: Other: Action observation therapy; Other: Exercise
- Exercise (Active Comparator): Strengthening and stretching exercises for hip and knee muscles, balance and proprioceptive exercises
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Action observation therapy — The normal human movement will be recorded and than the patients will be watched them.
  Arms: Action observation therapy and exercise
Other: Exercise — Strengthening and stretching exercise programme focuses on hip and knee muscles

SUMMARY:
The investigators aim to explore the effects of action observation therapy on pain and brain hemodynamics in patients with knee osteoarthritis. This study will create a new perspective to understand the physiology of pain, by applying painful stimulation during the neuroimaging system which has attracted much interest in the literature in recent years, and will shed light on the studies that can be done in this regard. Participants' pain level will be assessed using Visual Analog Scale and pressure algometer. Also joint range of motion in the initial assessments will be measured by electro-goniometer, muscle strength assessment by JTech hand dynamometer at appropriate evaluation positions. Fear of movement of individuals will be assessed via Tampa Kinesiophobia Scale and functional levels will be assessed via Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Timed Up and Go Test. Functional near infrared spectroscopy (fNIRS) will be used for evaluation of brain hemodynamics. The first group, will receive exercises with action observation therapy; and the second group will receive only exercises. The exercise programme will be administered under physiotherapist supervision for three days a week for six weeks. The evaluations will be repeated at the beginning of the study and at the end of the sixth week. Data obtained from the study will be analyzed using appropriate statistical methods.

DETAILED DESCRIPTION:
Osteoarthritic joint has pathological changes such as damage of joint cartilage tissue, thickening of the subchondral bone, osteophyte formation, inflammation of synovium at different levels, degeneration of ligaments and meniscal structures and hypertrophy of joint capsule. Pain is the most common symptom in osteoarthritic patients and the ongoing pain effects quality of life and physical functions of them negatively. At the same time, decrease in joint range of motion, muscle strength loss and decline in functional level may go along with pain. In recent years, studies that relate chronic pain to neuroplasticity have demonstrated changes in the structure, function and somatotopic organization of the primary motor and sensory cortex of osteoarthritis patients with chronic pain. In addition to this, osteoarthritis studies showed that the pain does not originate solely from joint problems; the central nervous system is also responsible for the formation of pain sensation. Changes in the cortical sensorimotor areas include sensory disturbances, perceptual problems (differentiation of body image), and motor influences, and these changes are associated with severity and duration of pain. It is reported that approaches targeting cortical reorganization resulted in decreased pain and increased function. Action observation therapy is a method which activates mirror neurons and is applied to learn a specific motor skill, facilitate motor learning and decrease the pain level of the extremities. It is anticipated that action observation therapy may differentiate perception of pain by altering cortical activity and thus altered motor cortical activity may play an active role in reducing pain by modulating pain-related neural networks.

The investigators aim to explore the effects of action observation therapy on pain and brain hemodynamics in patients with knee osteoarthritis. This study will create a new perspective to understand the physiology of pain, by applying painful stimulation during the neuroimaging system which has attracted much interest in the literature in recent years, and will shed light on the studies that can be done in this regard. Participants' pain level will be assessed using Visual Analog Scale and pressure algometer. Also joint range of motion in the initial assessments will be measured by electro-goniometer, muscle strength assessment by JTech hand dynamometer at appropriate evaluation positions.Fear of movement of individuals will be assessed via Tampa Kinesiophobia Scale and functional levels will be assessed via Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Timed Up and Go Test. Functional near infrared spectroscopy (fNIRS) will be used for evaluation of brain hemodynamics. The first group, will receive exercises with action observation therapy; and the second group will receive only exercises. The exercise programme will be administered under physiotherapist supervision for three days a week for six weeks. The evaluations will be repeated at the beginning of the study and at the end of the sixth week. Data obtained from the study will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* MMSE>21
* Chronic knee pain (VAS score>5)
* Right dominant
* Unilateral knee pain

Exclusion Criteria:

* Pain characteristics such as the presence of a rheumatologic disease other than knee osteoarthritis, lumbar radiculopathy, systemic inflammatory disease, diabetic neuropathy, problems similar to knee osteoarthritis,
* Hearing or vision problems,
* Injection therapy involving the knee region within the last 6 months,
* Surgical operation involving the knee region
* Psychiatric problems and anti-depressant usage

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Change in brain activation in dorsolateral prefrontal cortex as assessed by fNIRS monitoring (measure of hemodynamic response function) | 6 weeks
  In order to assess the brain hemodynamics during the painful and non painful stimulations of patients functional near infrared spectroscopy (NIRX Medical Technologies NIRScout) will be used. This neuroimaging method will be applied with 16 detector and 16 source which implanted via a cap. Firstly, the patients' pain pressure threshold level at knee region will be determined, then this value will be considered as painful stimulation. For non-painful stimulation 5 N will be applied to the patient. Hemodynamic responses will be evaluated according to the cortical areas (prefrontal cortex, premotor and supplementary motor cortex, primer motor cortex, primer somatosensory cortex)
Pain Level | 6 weeks
  Self reported pain intensity during the rest and the activity measured by Visual Analog Scale which presented as a 10 centimeter horizontal line and 0 means no pain, 10 means unbearable pain.
Pressure pain threshold | 6 weeks
  Algometer (dolorimeter) will be used to assess the pressure pain threshold, whereby the medial middle point of the knee and 2 cm lateral to the medial malleol.

SECONDARY OUTCOMES:
Kinesiophobia | 6 weeks
  Tampa Kinesiophobia Scale will be used to assess the fear of movement. It is a 17-item self report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury. The total score ranges between 17 and 68. A high value on the TSK indicates a high degree of kinesiophobia.
Western Ontario and Mcmaster Universities Osteoarthritis Index | 6 weeks
  WOMAC is used to assess pain, stiffness, and physical function in patients with knee osteoarthritis. Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing Stiffness (2 items): after first waking and later in the day Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.
Muscle strength | 6 weeks
  Hand-held dynamometer will be used to evaluate knee and hip muscles' strength.
Range of motion | 6 weeks
  Knee range of motion will be evaluated by digital goniometer. Knee flexion, knee extension, ankle dorsi and plantar flexion will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Özgül Öztürk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No